CLINICAL TRIAL: NCT04140253
Title: A Randomized-Intervention, Parallel, Multicentric Study to Evaluate Duloxetine and Innovative Pelvic Floor Muscle Training in Women With Uncomplicated Stress Urinary Incontinence - The DULOXING Study
Brief Title: Evaluation of Duloxetine and Innovative Pelvic Floor Muscle Training in Women With Stress Urinary Incontinence
Acronym: DULOXING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Comenius University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24012019
Record Dates: First submitted 2019-10-22; First posted 2019-10-25 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Stress Urinary Incontinence in Women
Keywords: Stress urinary incontinence; Pelvic floor muscle training
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Duloxetine treatment (Active Comparator): Peroral treatment with duloxetine at a dose of 40 mg twice a day
  Interventions: Behavioral: Pelvic floor muscle training (PFMT) with lumbopelvic stabilization
- Standard Duloxetine treatment with PFMT (Experimental): Peroral treatment with duloxetine at a dose of 40 mg twice a day. Pelvic floor muscle training (PFMT) with lumbopelvic stabilization.
  Interventions: Behavioral: Pelvic floor muscle training (PFMT) with lumbopelvic stabilization

INTERVENTIONS:
Behavioral: Pelvic floor muscle training (PFMT) with lumbopelvic stabilization — Pelvic floor muscle training (PFMT) with lumbopelvic stabilization.
  1. Educating of probands about anatomy, physiology, and pelvic floor muscles functions
  2. Training of pelvic floor muscles in different position
  3. Training of pelvic floor muscles with lumbopelvic stabilization
  Exercise 5 times a week for 20-30 minutes a day, after initial training with a physiotherapist.

SUMMARY:
This study will evaluate the safety, tolerability and efficacy of duloxetine and pelvic floor muscle training in women who suffer from stress urinary incontinence

DETAILED DESCRIPTION:
This is a randomized-intervention, parallel, multicentric study which will evaluate the safety, tolerability and efficacy of oral duloxetine and innovative pelvic floor muscle training to woman suffering from stress urinary incontinence

ELIGIBILITY:
Inclusion Criteria:

* Woman's willing to provide written informed consent
* Women over 18 years that experience uncomplicated stress urinary incontinence
* Score of the International Consultation on Urinary Incontinence Questionnaire ≥ 14 points
* Symptoms of urinary incontinence for at least 3 consecutive months
* Have at least seven urinary incontinence episodes per week
* Degree of pelvic organ prolapse ≤ 2 stage
* Willingness to accept the randomization process and fully participate in tests

Exclusion Criteria:

* Recent use of any pharmacologic agent used to treat symptoms of urinary incontinence in the past six months
* History of anti-incontinence surgery in the past 12 months
* Use of onabotulinumtoxinA for the treatment of urinary incontinence in the past 12 months
* History of pelvic prolapse repair or urethral surgery in the past 12 months
* History of pelvic floor muscle training in the past 12 months
* History of interstitial cystitis or bladder-related pain
* Chronic severe constipation
* Clinically significant renal or hepatic impairment
* Clinically significant heart impairment
* Pregnant woman, lactating, or actively trying to become pregnant
* Non-compliance with limitation of duloxetine treatment for mixed urinary incontinence
* Positive urinary tract infection
* Use of rehabilitation aids (pessary, urethral plugs, vaginal beads, etc.)
* Use of antidepressant therapy
* Insufficient understanding of pelvic floor exercises and/or omitting exercises
* Participation in any clinical study in the past six months

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — woman with stress urinary incontinence
Enrollment: 158 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Change in incontinence episode frequency | over 12 weeks of treatment
  The investigators will compare change in incontinence episode frequency in the combined duloxetine and pelvic floor muscle training to duloxetine treatment alone

SECONDARY OUTCOMES:
Change in incontinence quality of life according to Incontinence Quality of Life scale (I-QoL) | over 12 weeks of treatment
  The investigators will compare change in incontinence quality of life in the combined duloxetine and pelvic floor muscle training to duloxetine treatment alone. 0 = worst quality of life, 100 = best quality of life.
Change in Patient Global Impression of Improvement (PGI-I score) | over 12 weeks of treatment
  To examine change in Patient Global Impression of Improvement in the combined duloxetine and pelvic floor muscle training to duloxetine treatment alone . 1 = much better. 7 = definitely worse.
Incidence of adverse events | over 12 weeks of treatment
  To examine incidence of adverse events in the combined duloxetine and pelvic floor muscle training to duloxetine treatment alone

CONTACTS AND LOCATIONS:
Locations (1):
- Jessenius Faculty of Medicine in Martin, Comenius University in Bratislava, Martin, Slovakia

IPD SHARING:
Plan to Share IPD: No
After study completion

REFERENCES:
- [Derived] Hagovska M, Svihra J, Breza J Jr, Dubravicky J, Vargovcak M. A randomized, intervention parallel multicentre study to evaluate duloxetine and innovative pelvic floor muscle training in women with uncomplicated stress urinary incontinence-the DULOXING study. Int Urogynecol J. 2021 Jan;32(1):193-201. doi: 10.1007/s00192-020-04516-w. Epub 2020 Aug 27. PMID 32852574
- [Derived] Hagovska M, Svihra J. Evaluation of duloxetine and innovative pelvic floor muscle training in women with stress urinary incontinence (DULOXING): Study protocol clinical trial (SPIRIT Compliant). Medicine (Baltimore). 2020 Feb;99(6):e18834. doi: 10.1097/MD.0000000000018834. PMID 32028393